CLINICAL TRIAL: NCT04167761
Title: Ertugliflozin: Cardioprotective Effects on Epicardial Fat
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tracey McLaughlin, Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 52647
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Type 2 Diabetes; Insulin Resistance
Keywords: Epicardial Adipose Tissue; SGLT2 Inhibitor
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — ertugliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: in vitro experimental study with treated and control tissue samples
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ertugliflozin (treated tissue) (Experimental): Adipose tissue samples collected from participants were treated with Ertugliflozin at a concentration of 25 µM in vitro. Tissue samples were incubated with Ertugliflozin to evaluate its effects on lipolysis, inflammation, and gene expression in epicardial, pericardial, and subcutaneous adipose tissues
  Interventions: Drug: Ertugliflozin

INTERVENTIONS:
Drug: Ertugliflozin — Adipose tissue samples collected from participants were treated with Ertugliflozin at a concentration of 25 µM in vitro. This treatment was applied in a laboratory setting to assess the effects of Ertugliflozin on lipolysis, inflammatory cytokine release, and gene expression in epicardial, pericardial, and subcutaneous adipose tissue
  Other Names: SGLT2 inhibitor

SUMMARY:
The purpose of this study is to learn if Sodium-Glucose Cotransporter 2 inhibitor (SGLT2i) medications enhance beneficial properties of epicardial adipose tissue including metabolic flexibility, insulin sensitivity, decreased cell size and reduced inflammation.

ELIGIBILITY:
Inclusion Criteria:

* patient at Stanford Cardiovascular Surgery clinic who is scheduled for cardiac bypass surgery or vascular surgery
* history of Diabetes Mellitus Type 2 currently diet controlled, or on metformin or dpp4 inhibitors

Exclusion Criteria:

* allergy or intolerance to interventional medication
* currently taking insulin, glp-1 inhibitors, or sulfonylureas

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of isoproterenol-stimulated lipolysis to measure metabolic flexibility in epicardial adipose tissue samples. | Time to collect tissue collected during surgery (up to 15 minutes)
  Analysis will be performed using Lipolysis Colorimetric Assay and measured by glycerol content on standard curve. Indirect effects of SGLT2i in vivo in epicardial adipose tissue will be compared to Glipizide by measuring rate of lipolysis, or breakdown of adipose in to free fatty acids.

SECONDARY OUTCOMES:
Average insulin mediated glucose uptake (IMGU) to measure insulin sensitivity in epicardial adipose tissue samples. | Time to collect tissue collected during surgery (up to 15 minutes)
  Mature adipocytes will be isolated, cultured, and treated with 2-NBDG, a fluorescently-labeled deoxyglucose analog, as a probe for the detection of glucose uptake measured by excitation/emission of florescence in the mature cells.
Characterization of the inflammatory cytokine expression profile in epicardial adipose tissue samples. | Time to collect tissue collected during surgery (up to 15 minutes)
  Analysis will be performed using Luminex to measure levels of inflammatory cytokines on the human adipocyte panel.
Distribution of adipose cell size in epicardial tissue. | Time to collect tissue collected during surgery (up to 15 minutes)
  After tissue collection and osmium fixation, adipose cell size will be determined by Beckman Coulter Multisizer III, and described via a mathematical model to estimate peak diameter, fat storage capacity, size variability, and % small cells.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT04167761/Prot_SAP_000.pdf